CLINICAL TRIAL: NCT00300183
Title: Evaluation of an Outreach and Intervention Program to Reach HIV- Positive Persons Living in Bronx, NY Single Room Occupancy Hotels
Brief Title: Evaluation of an HIV Outreach Program
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); CitiWide Harm Reduction (Other)
Responsible Party: Sponsor
Other Study IDs: 02-02-038; 2H97 HA 00247-03-02 (Other Grant/Funding Number: Health Resources and Services Administration (HRSA))
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV; health services accessibility; health services research; homeless; social support; AIDS; substance abuse; mental health; quality of life; outreach; harm reduction
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Psychological Well-Being; Harm Reduction

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study evaluates outreach to HIV-infected people living in unstable housing in New York City who are new to CitiWide Harm Reduction. One hundred and fifty people are interviewed every 6 months, and their medical records are reviewed every 6 months for a total of 18 months. The study examines how outreach, case management, housing, drug use, mental health, and quality of life are related to people's ability to get into and stay in medical care.

DETAILED DESCRIPTION:
The study is a prospective cohort study in which 150 newly enrolled HIV-infected participants of CitiWide Harm Reduction are followed for 18 months to assess HIV-related health outcomes. Data elements include (1) face-to-face interviews focusing on housing, HIV disease severity, utilization of health care services, utilization of non-medical services, substance use, mental health, and quality of life; (2) medical chart information focusing on CD4 count, viral load, and HIV primary care visits; and (3) outreach services. The study hypothesis is that involvement with CitiWide Harm Reduction will improve HIV-related health care utilization and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected, living in one of 15 single room occupancy hotels served by CitiWide Harm Reduction, new to CitiWide Harm Reduction, at least 18 years of age, English or Spanish speaking

Exclusion Criteria:

* HIV-negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-10 (Actual); Primary Completion 2005-07-31 (Actual); Study Completion 2005-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chinazo O Cunningham, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States